CLINICAL TRIAL: NCT03346967
Title: Evaluation of Autologous Adipose Derived Mesenchymal Stem Cells (AD-MSCs) Therapy on Sexual Hormone Deficiency in the Middle-aged Patients: an Open-label, Single-group Clinical Trial
Brief Title: Outcomes of Adipose Derived Mesenchymal Stem Cells on Sexual Hormone Deficiency
Acronym: MSCSHD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VinmecRISCGT72
Record Dates: First submitted 2017-11-14; First posted 2017-11-20 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Hormone Deficiency
Keywords: AD mesenchymal stem cells;sexual hormone deficiency

STUDY DESIGN:
Intervention Model Description: 30 patients with sexual hormone deficiency will be injected AD-MSCs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stem cell Administration for female patients (Experimental): Single Intravenous Administration of Autologous Adipose-derived Mesenchymal Stem Cells with Dosage at 1 million cells per body-weight kilogram for female patients
  Interventions: Combination Product: adipose-derived mesenchymal stem cells
- Stem cell Administration for male patients (Experimental): Single Intravenous Administration of Autologous Adipose-derived Mesenchymal Stem Cells with Dosage at 1 million cells per body-weight kilogram for male patients
  Interventions: Combination Product: adipose-derived mesenchymal stem cells

INTERVENTIONS:
Combination Product: adipose-derived mesenchymal stem cells — Collect adipose-derived mesenchymal stem cells from the patients. Adipose-derived mesenchymal stem cells will be isolated, expanded and characterized in vitro under the GMP- grade procedure

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of adipose derived mesenchymal stem cells (AD-MSCs) therapy on sexual hormone deficiency in the middle-aged patients

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficiency of adipose-derived mesenchymal stem cells in 30 patients with sexual hormone deficiency at Vinmec International Hospital, Hanoi, Vietnam

ELIGIBILITY:
Inclusion Criteria:

* Age: 35 years to 70 years (Male) and from 35 years to menopause age (Female)
* Male: decrease in libido, decrease in intercourse frequency, erectile dysfunction, Difficulty in concentration, testosterone level ≤ 12 nMol/dL
* Female: reduced or absent menstruation after radiation exposure or chemotherapy; Hot flushes, excessive sweating, and anxiety, together with other symptoms associated with the menopause, AMH level ≤ 2 ng/ml and/or FSH level ≥ 10 mIU/ml.
* Patients signed the informed consent form

Exclusion Criteria:

* Surgery removal of endocrine glands
* Abnormalities in the endrocrine glands
* Hormone deficiency due to diabetes and other metabolic disorders
* Active autoimmune diseases
* Current usage of immunosuppressive drugs
* Coagulation disorders
* Allergy to anesthetic agents
* Severe health conditions such as cancer, failure of heart, lung, liver or kidney
* Active infections

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — * 40 years to 65 years (Male) and from 40 years to menopause age (Female)
  * Male: decrease in libido, decrease in intercourse frequency, erectile dysfunction, Difficulty in concentration, testosterone level ≤ 12 nMol/dL
  * Female: reduced or absent menstruation after radiation exposure or chemotherapy; Hot flushes, excessive sweating, and anxiety, together with other symptoms associated with the menopause, AMH level ≤ 2 ng/ml and/or FSH level ≥ 10 mIU/ml.
Enrollment: 30 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Serum levels of follicle-stimulating hormone (FSH), Anti-Mullerian Hormone (AMH) and estradiol (E2) for female and testosterone level for male | up to the 12-month period following treatment
  Comparison between Serum levels of follicle-stimulating hormone (FSH), Anti-Mullerian Hormone (AMH) and estradiol (E2) for female and testosterone level for male at pre and post AD-MSCs therapy

CONTACTS AND LOCATIONS:
Overall Officials: Liem Nguyen, PhD, Principal Investigator — Vinmec Healthcare System
Locations (1):
- Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reed-Maldonado AB, Lue TF. The Current Status of Stem-Cell Therapy in Erectile Dysfunction: A Review. World J Mens Health. 2016 Dec;34(3):155-164. doi: 10.5534/wjmh.2016.34.3.155. Epub 2016 Dec 22. PMID 28053944
- [Result] Haahr MK, Jensen CH, Toyserkani NM, Andersen DC, Damkier P, Sorensen JA, Lund L, Sheikh SP. Safety and Potential Effect of a Single Intracavernous Injection of Autologous Adipose-Derived Regenerative Cells in Patients with Erectile Dysfunction Following Radical Prostatectomy: An Open-Label Phase I Clinical Trial. EBioMedicine. 2016 Jan 19;5:204-10. doi: 10.1016/j.ebiom.2016.01.024. eCollection 2016 Mar. PMID 27077129
- [Result] Charles-de-Sa L, Gontijo-de-Amorim NF, Maeda Takiya C, Borojevic R, Benati D, Bernardi P, Sbarbati A, Rigotti G. Antiaging treatment of the facial skin by fat graft and adipose-derived stem cells. Plast Reconstr Surg. 2015 Apr;135(4):999-1009. doi: 10.1097/PRS.0000000000001123. PMID 25811565
- [Derived] Nguyen Thanh L, Dam PTM, Nguyen HP, Nguyen TT, To HM, Nguyen HB, Luu NA, Hoang DM. Can Autologous Adipose-Derived Mesenchymal Stem Cell Transplantation Improve Sexual Function in People with Sexual Functional Deficiency? Stem Cell Rev Rep. 2021 Dec;17(6):2153-2163. doi: 10.1007/s12015-021-10196-w. Epub 2021 Jun 15. PMID 34129158